CLINICAL TRIAL: NCT01492465
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Ascending Single Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AMG 876 in Subjects With Type 2 Diabetes
Brief Title: Single Ascending Dose Trial in Patients With Type 2 Diabetes
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Decision by Sponsor
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20100015
Record Dates: First submitted 2011-09-28; First posted 2011-12-15 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Diabetes Mellitus
Keywords: Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- AMG 876 (Active Comparator)
  Interventions: Drug: AMG 876
- Placebo (Placebo Comparator)
  Interventions: Drug: AMG 876

INTERVENTIONS:
Drug: AMG 876 — Ascending single doses of study drug administered SC, with one cohort administered IV

SUMMARY:
The purpose of this study is to determine whether AMG 876 is safe and well tolerated in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided written informed consent
* Men and women between the ages of 18 and 65, inclusive at the time of randomization
* Women must be of documented non-reproductive potential (ie, postmenopausal [see definition below]; OR history of hysterectomy; OR history of bilateral tubal ligation; OR history of bilateral oophorectomy).
* Diagnosed with type 2 diabetes
* HbA1c ≥ 6.5% and ≤ 10%
* Fasting C-peptide value ≥ 0.8 ng/mL
* Men must agree for the duration of the study and continuing for 4 weeks after the dose of study drug, to practice a highly effective method of birth control. Highly effective methods of birth control include sexual abstinence, vasectomy or a condom with spermicide (men) in combination with either barrier methods, hormonal birth control or IUD (women).
* Men must agree to not donate sperm for the duration of the study and continuing for 4 weeks after the dose of study drug.
* Body mass index between ≥ 25.0 kg/m2 and ≤ 40.0 kg/m2 at screening
* Negative screening test for alcohol and potential drugs of abuse at screening and day -2, unless medication is prescribed by a physician and approved by the principal investigator and Amgen medical monitor

Exclusion Criteria:

* Men with partners who are pregnant at the time of screening or men with partners who plan to become pregnant during the study
* Women who are pregnant or breastfeeding History or evidence of a clinically significant disorder, condition or disease that, in the opinion of the principal investigator or Amgen medical monitor would pose a risk to subject safety or interfere with the study evaluation, procedures or completion
* Evidence or history at screening of diabetic complications with significant end-organ damage, eg, proliferative retinopathy and/or macular edema, creatinine clearance < 60 mL/min/1.73m2 (calculated using the Modification of Diet in Renal Disease formula), or macroalbuminuria (ie, ≥ +1 proteinuria on urinalysis), diabetic neuropathy complicated by neuropathic ulcers, or severe autonomic neuropathy with gastroparesis, chronic diarrhea, or hypoglycemic unawareness
* Significant cardiac disease, including but not limited to evidence or history of coronary artery disease, unstable angina, congestive heart failure, known arrhythmias of ventricular etiology, unexplained syncope or syncope/seizures related to arrhythmia
* Positive for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (Hbs Ag), or hepatitis C virus antibodies
* An unstable medical condition, defined as having been hospitalized within 28 days before day -1, major surgery within 6 months before day -1, or otherwise unstable in the judgment of the investigator (eg, risk of complications or adverse events unrelated to study participation)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2011-11; Primary Completion 2012-07 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Subject incidence of treatment-emergent adverse events | 29 days
  Physical examinations, vitals, clinical laboratories, and ECGs
Safety laboratory analytes, vital signs, and ECGs | 29 days
  laboratory analytes, vital signs, and ECGs
Subject incidence of anti-AMG 876 antibodies. | 29 days
  laboratories analytes

SECONDARY OUTCOMES:
AMG 876 serum PK parameters | 29 days
  Concentration-time profiles for AMG 876
Pharmacodynamic parameters: | 29 days
  Concentration of fasting glucose, insulin and c-peptide levels; Concentration-time profiles and AUC for metabolic parameters (eg, glucose, insulin, c-peptide, glucagon and free fatty acid concentrations) following a mixed meal tolerance test; Lipid levels (ie, total cholesterol, LDL, HDL, and triglycerides); Body weight.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (3):
- United States (3):
  - Research Site, Omaha, Nebraska
  - Research Site, San Antonio, Texas
  - San Antonio, Texas

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com